CLINICAL TRIAL: NCT00419705
Title: NeuroThera® Effectiveness and Safety Trial - 2 (NEST-2) A Double Blind, Randomized, Controlled, Parallel Group, Multicenter, Pivotal Study to Assess the Safety and Effectiveness of the Treatment of Acute Ischemic Stroke With the NeuroThera® Laser System Within 24 Hours From Stroke Onset
Brief Title: Effectiveness and Safety Trial of a New Ischemic Stroke Treatment Within 24 Hours From Stroke Onset (NEST-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PhotoThera, Inc (Industry)
Responsible Party: Jackson Streeter, MD, PhotoThera, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTS-INT06-007
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Ischemic Stroke
Keywords: acute stroke; infrared laser therapy; clinical trial; safety; effectiveness
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Laser Therapy (Experimental)
  Interventions: Device: NeuroThera® Laser System
- Sham control procedure (Sham Comparator)
  Interventions: Device: NeuroThera® Laser System

INTERVENTIONS:
Device: NeuroThera® Laser System — Transcranial delivery of laser therapy or sham (no laser therapy) to the scalp

SUMMARY:
The purpose of this pivotal study is to demonstrate safety and effectiveness of the NeuroThera® Laser System (referred to hereafter as NTS) in the treatment of Subjects diagnosed with acute ischemic stroke. The initiation of NTS treatment must be feasible for each Subject within 24 hours of stroke onset.

DETAILED DESCRIPTION:
This study is a prospective, double blind, randomized, sham controlled, parallel group, multi-center study that will include enrollment of up to 660 Subjects. Subjects will be followed for 90 days post stroke onset. The primary effectiveness endpoint for this study will be the binary endpoint that defines success as a modified Rankin Scale (mRS) score of 0-2 and failure as an mRS score of 3-6 at 90 days or the last rating. The secondary effectiveness endpoint for this study will be the change in NIHSS score from baseline to 90 days or the last rating, analyzed across the full range of scores on the NIHSS. Tertiary effectiveness endpoints include: The 90-day binary endpoint, denoted as the 90-day bNIH score, based on the NIHSS score that defines a successful result as either (i) an improvement of 9 or more points on the NIHSS or (ii) a final NIHSS score of 0 or 1; the score on the mRS at 90 days or the last rating analyzed across the range of scores from 0 to 6 on the mRS scale, SIS-16 at 90 days; mortality at 30, 60 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Acute Ischemic Stroke within 24 hours
2. Clinical diagnosis of Acute Ischemic Stroke after exclusion of hemorrhage by a CT scan or susceptibility weighted MRI sequences
3. NIHSS ≥7 - ≤22

Exclusion Criteria:

1. >24hours from symptom onset to time of treatment
2. Evidence of intracranial, subdural, or subarachnoid hemorrhage
3. Clinical presentation of intracranial hemorrhage
4. Pre stroke ≥3 mRS
5. The presence of a brainstem or cerebellar stroke
6. Transient Ischemic Attack (TIA)
7. Seizure at stroke onset
8. Blood glucose >400 or <60
9. Sustained systolic BP >220mmHG < 80mmHG or diastolic >140mmHG <50mmHG
10. Septic embolus
11. CNS tumor (except asymptomatic meningioma)
12. Dermatologic condition of the scalp (e.g. Psoriasis)
13. Thrombolytic therapy
14. Head implant (e.g. Clipped aneurysm, Hakim valve)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Disability scale (mRS)score at 90 days; safety of the treatment procedure | at baseline, day 5, 30, 60 and 90 post treatment

SECONDARY OUTCOMES:
Functional neurological scale(NIHSS)over time | at baseline, Day 5, 30, 60 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Justin Zivin, MD, PhD, Study Chair — University of California San Diego, Department of Neurosciences; 9500 Gillman Drive; La Jolla, CA 92093
Locations (58):
- United States (51):
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Alta Bates Summit Medical Center, Berkeley, California
  - Scripps Encinitas Hospital, Encinitas, California
  - Grossmont Hospital, La Mesa, California
  - UCLA Medical Center, Los Angeles, California
  - Tri City Medical Center, Oceanside, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Sharp Healthcare, San Diego, California
  - Neurology Medical Group of Diablo Valley, Walnut Creek, California
  - Swedish Medical Center, Englewood, Colorado
  - The Stroke Center at Hartford Hospital, Hartford, Connecticut
  - North Broward Medical Center, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Naples Community Hospital, Naples, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Dekalb Medical Center, Decatur, Georgia
  - Dekalb Neurology Associates LLC, Decatur, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Intensive Care Unit, Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Benefis Healthcare East Campus, Great Falls, Montana
  - Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - UNC Health Care, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - The University Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Hospital, Portland, Oregon
  - Oregon Health & Science University - Oregon Stroke Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Charleston Area Medical Center (CAMC) General Hospital, Charleston, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Germany (4):
  - Neurologische Klinik des Universitatsklinikum Erlangen, Erlangen
  - Neurologische Klinik des Universitatsklinikum Heidelberg, Heidelberg
  - Klinik und Poliklinik fur Neurologic Leipzig, Leipzig
  - Neurologische Klinik und Poliklinik Westfalische Wilhelms Universitat, Münster
- Hospital Nacional "Dos de Mayo", Lima, Peru
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Sjukhuset i Lidkoping, Lidköping

REFERENCES:
- [Result] Zivin JA, Albers GW, Bornstein N, Chippendale T, Dahlof B, Devlin T, Fisher M, Hacke W, Holt W, Ilic S, Kasner S, Lew R, Nash M, Perez J, Rymer M, Schellinger P, Schneider D, Schwab S, Veltkamp R, Walker M, Streeter J; NeuroThera Effectiveness and Safety Trial-2 Investigators. Effectiveness and safety of transcranial laser therapy for acute ischemic stroke. Stroke. 2009 Apr;40(4):1359-64. doi: 10.1161/STROKEAHA.109.547547. Epub 2009 Feb 20. PMID 19233936